CLINICAL TRIAL: NCT04163887
Title: Effect of the Laparoscopic Approach in Reducing Postoperative Severe Complications Following Hepatectomy for Colorectal Liver Metastases: Prospective, Randomized, Controlled Study
Brief Title: Effect of the Laparoscopic Approach in Reducing Postoperative Severe Complications Following Hepatectomy for Colorectal Liver Metastases
Acronym: METALAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Ministry of Health, France (Other Government); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIG-03-2019
Record Dates: First submitted 2019-10-21; First posted 2019-11-15 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Liver Metastasis Colon Cancer; Postoperative Complications
Keywords: Liver resection; Laparoscopy
MeSH Terms: conditions — Postoperative Complications | interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: Prospective multicenter, open-label and pragmatic, controlled randomized (minimization procedure) superiority trial in 2 parallel groups comparing the rates of 90 days postoperative complications between patients undergoing laparoscopic and open liver resection for colorectal liver metastases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic liver resection (Other): Laparoscopy allows some surgical procedures to be performed through small incisions that enable the operator to access the abdominal cavity, often at the pubic area, and surgical instruments are introduced through these small incisions. This technique avoids large abdominal incisions and significantly reduces the duration of hospitalization.
  Interventions: Procedure: hepatectomy
- open liver resection (Other): standard of care
  Interventions: Procedure: hepatectomy

INTERVENTIONS:
Procedure: hepatectomy — Resection colorectal liver metastases using a laparoscopic approach or an open approach.

SUMMARY:
The objective of this study is to demonstrate the superiority of the laparoscopic approach over the open approach in the resection of colorectal liver metastases, by examining the reduction of postoperative complications (including mortality), measured using the Comprehensive Complication Index (CCI) within 90 days of the procedure or regardless of the date during the hospital stay.

DETAILED DESCRIPTION:
While laparotomy is still the standard approach of resectable colorectal liver mestastases, its associated morbidity remains non-negligible with reported mortality and complications rates ranging from 2 to 8% and 30 to 70%, respectively (1). Besides the underlying liver disease together with the comorbidities of the patients, this high morbidity is also related to the type of surgical approach. Since less than 15% of liver resections are currently performed using the laparoscopic approach in France, a trial showing the superiority of the laparoscopic approach in comparison to the open approach for patients with colorectal liver metastases qualifying for both approaches would allow improving management of patients, reducing the length of stay, maybe decreasing the global cost and changing current practices on a national scale.

In order to demonstrate the superiority of the laparoscopic approach over the laparotomy approach, patients with colorectal hepatic metastasis will be randomly assigned to either the laparoscopy or laparotomy groups. Post-operative complications (including mortality) will be measured using the Comprehensive Complication Index (CCI) within 90 days postoperatively or at any time during hospitalization. The participation time for each patient in the study is 3 years, the patient will be followed at 1, 3, 6, 9, 9, 12, 15, 18, 21, 24, 30 and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with colorectal liver metastases requiring liver resection ± concomitant radiofrequency ablation.
* Qualifying for both a laparoscopic approach and an open approach.
* Informed written consent.
* Affiliated to health insurance regimen.

Exclusion Criteria:

* Hybrid liver resection (including both laparoscopic and open resection).
* Liver resection requiring an associated vascular or biliary reconstruction.
* Contraindication to surgery.
* Contraindication to laparoscopy (pneumoperitoneum).
* ASA (American Society of Anesthesiologists) score IV or V or life expectancy < 3 months.
* Poor comprehension of French language or cognitive impairment
* Pregnancy or breastfeeding.
* Patient under guardianship or unable to give consent
* People particularly protected by French law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-04-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Rate of overall complications using the comprehensive complication Index (CCI) | Within 90 days postoperatively or at any time during hospitalization.
  CCI is calculated using the burden of postoperative complications weighted with a measure of the severity according to the widely accepted Dindo-Clavien classification of postoperative complications and a dedicated CCI calculator.

SECONDARY OUTCOMES:
Proportion of patients presenting severe postoperative complications | Within 90 days postoperatively or at any time during hospitalization.
  Proportion of patients presenting severe postoperative complications rate as defined by the Clavien-Dindo classification ≥ grade 3 (including mortality) between patients treated with laparoscopic liver resection and those treated with open liver surgery
Rate of conversion from laparoscopy liver resection to open liver surgery | during surgery.
  Conversion is defined as the requirement for laparotomy at any time of the procedure with the exception of the extraction of the resected specimen. Specific data regarding conversion will be noticed from the operative reports. These included the reasons for conversion, the timing of conversion and the type of conversion.
Length of hospital stay | Within 90 days postoperatively or at any time during hospitalization.
  Length of hospital stay and occurrence of unplanned readmission after discharge,assessed by hospitalization reports
Delay of recovery before resuming professional activities. | Within 90 days postoperatively
  Delay of recovery before resuming professional activities assessed by PQRS (Postoperative Quality Recovery Scale) including nociceptive domain, emotional domain, cognition domain and day-to-day activities at D-1, D1, D7, D30 and D90.
Postoperative quality of life using quality of life questionnaries. | At the inclusion (before surgery), at 1 month postintervention, 3 months, 6 months and then every 6 months during 3 years.
  Patient-reported outcome measures were assessed with the validated European Organisation for Research and Treatment of Cancer (EORTC) score questionnaire, EORTC Quality of Life Questionnaire (QLQ) -C30 (version 3.0), and the module dedicated to colorectal liver metastases (EORTC QLQ-LMC21). EQ5D-5L is a standardised measure of health status that provides a simple descriptive profile and a single index value suitable for the economic evaluation of health. It will be used to calculate the QALYs of each enrolled patient, by valuing health.
Health economics analysis | During the full participation period (3 years).
  A cost-effectiveness study will be performed and completed by a cost-utility analysis to identify the efficient therapeutic strategy (laparoscopic approach) ompared to the reference (open surgery).
  Only direct costs will be considered for treatments, management of side effects, medical transports, rehabilitation procedures and medical consultations.
  Out of hospital resources are valued from the Social Health Insurance (SHI) tariffs and hospital stays the Diagnosis-Related group (DRG) tariff taking into account additional daily fixed prices for ICU stay, if any.
Oncologic quality of the resection using the pathological report. | During surgery
  Mean surgical margin widths (in millimeters). Percentages of microscopically complete (R0), microscopically incomplete (R1) and macroscopically incomplete (R2) resections as stated in the pathological report.
Disease-free and overall survival at 3 years. | During the full participation period (3 years).
  1. Percentage of patients with intrahepatic or extrahepatic recurrence three years after the operation.
  2. Median disease-free survival time (in months).
  3. Percentage of patients who died at 1, 2 and 3 years after the procedure.
  4. Median overall survival time (in months).

CONTACTS AND LOCATIONS:
Overall Officials: David FUKS, PR, Study Chair — Institut Mutualiste Montsouris
Locations (21):
- France (21):
  - CHU Amiens Picardie, Amiens
  - Hôpital Côte de Nacre - Chu Caen, Caen
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - CHU Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hôpital Claude Huriez, Lille
  - HCL - Hôpital Croix Rousse, Lyon
  - CHU de Marseille Hôpital de Timone, Marseille
  - l'Institut Paoli Calmettes, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy - Hôpitaux Brabois, Nancy
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Cochin, Paris
  - Hôpital La pitié Salpêtrière, Paris
  - CHU de Reims, Reims
  - Hôpital Charles Nicolle, Rouen
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU Rangueil, Toulouse
  - Hôpital Trousseau, Tours
  - Hôpital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2015. CA Cancer J Clin. 2015 Jan-Feb;65(1):5-29. doi: 10.3322/caac.21254. Epub 2015 Jan 5. PMID 25559415
- [Background] Manfredi S, Lepage C, Hatem C, Coatmeur O, Faivre J, Bouvier AM. Epidemiology and management of liver metastases from colorectal cancer. Ann Surg. 2006 Aug;244(2):254-9. doi: 10.1097/01.sla.0000217629.94941.cf. PMID 16858188
- [Background] Power DG, Kemeny NE. Role of adjuvant therapy after resection of colorectal cancer liver metastases. J Clin Oncol. 2010 May 1;28(13):2300-9. doi: 10.1200/JCO.2009.26.9340. Epub 2010 Apr 5. PMID 20368552
- [Background] Komatsu S, Scatton O, Goumard C, Sepulveda A, Brustia R, Perdigao F, Soubrane O. Development Process and Technical Aspects of Laparoscopic Hepatectomy: Learning Curve Based on 15 Years of Experience. J Am Coll Surg. 2017 May;224(5):841-850. doi: 10.1016/j.jamcollsurg.2016.12.037. Epub 2017 Jan 20. PMID 28111192
- [Background] Fuks D, Cauchy F, Fteriche S, Nomi T, Schwarz L, Dokmak S, Scatton O, Fusco G, Belghiti J, Gayet B, Soubrane O. Laparoscopy Decreases Pulmonary Complications in Patients Undergoing Major Liver Resection: A Propensity Score Analysis. Ann Surg. 2016 Feb;263(2):353-61. doi: 10.1097/SLA.0000000000001140. PMID 25607769
- [Background] Nomi T, Fuks D, Ogiso S, Nakajima Y, Louvet C, Gayet B. Second and Third Laparoscopic Liver Resection for Patients With Recurrent Colorectal Liver Metastases. Ann Surg. 2016 May;263(5):e68-72. doi: 10.1097/SLA.0000000000001528. No abstract available. PMID 26641255
- [Background] Ciria R, Cherqui D, Geller DA, Briceno J, Wakabayashi G. Comparative Short-term Benefits of Laparoscopic Liver Resection: 9000 Cases and Climbing. Ann Surg. 2016 Apr;263(4):761-77. doi: 10.1097/SLA.0000000000001413. PMID 26700223
- [Background] Hallet J, Sa Cunha A, Cherqui D, Gayet B, Goere D, Bachellier P, Laurent A, Fuks D, Navarro F, Pessaux P; French Colorectal Liver Metastases Working Group, Association Francaise de Chirurgie. Laparoscopic Compared to Open Repeat Hepatectomy for Colorectal Liver Metastases: a Multi-institutional Propensity-Matched Analysis of Short- and Long-Term Outcomes. World J Surg. 2017 Dec;41(12):3189-3198. doi: 10.1007/s00268-017-4119-z. PMID 28717911
- [Background] Fretland AA, Dagenborg VJ, Bjornelv GMW, Kazaryan AM, Kristiansen R, Fagerland MW, Hausken J, Tonnessen TI, Abildgaard A, Barkhatov L, Yaqub S, Rosok BI, Bjornbeth BA, Andersen MH, Flatmark K, Aas E, Edwin B. Laparoscopic Versus Open Resection for Colorectal Liver Metastases: The OSLO-COMET Randomized Controlled Trial. Ann Surg. 2018 Feb;267(2):199-207. doi: 10.1097/SLA.0000000000002353. PMID 28657937
- [Background] Gilg S, Sparrelid E, Isaksson B, Lundell L, Nowak G, Stromberg C. Mortality-related risk factors and long-term survival after 4460 liver resections in Sweden-a population-based study. Langenbecks Arch Surg. 2017 Feb;402(1):105-113. doi: 10.1007/s00423-016-1512-2. Epub 2016 Oct 1. PMID 27695941
- [Background] Cannon RM, Scoggins CR, Callender GG, McMasters KM, Martin RC 2nd. Laparoscopic versus open resection of hepatic colorectal metastases. Surgery. 2012 Oct;152(4):567-73; discussion 573-4. doi: 10.1016/j.surg.2012.07.013. Epub 2012 Sep 1. PMID 22943842
- [Background] Beppu T, Wakabayashi G, Hasegawa K, Gotohda N, Mizuguchi T, Takahashi Y, Hirokawa F, Taniai N, Watanabe M, Katou M, Nagano H, Honda G, Baba H, Kokudo N, Konishi M, Hirata K, Yamamoto M, Uchiyama K, Uchida E, Kusachi S, Kubota K, Mori M, Takahashi K, Kikuchi K, Miyata H, Takahara T, Nakamura M, Kaneko H, Yamaue H, Miyazaki M, Takada T. Long-term and perioperative outcomes of laparoscopic versus open liver resection for colorectal liver metastases with propensity score matching: a multi-institutional Japanese study. J Hepatobiliary Pancreat Sci. 2015 Oct;22(10):711-20. doi: 10.1002/jhbp.261. Epub 2015 May 21. PMID 25902703
- [Background] Adam R, Pascal G, Azoulay D, Tanaka K, Castaing D, Bismuth H. Liver resection for colorectal metastases: the third hepatectomy. Ann Surg. 2003 Dec;238(6):871-83; discussion 883-4. doi: 10.1097/01.sla.0000098112.04758.4e. PMID 14631224
- [Background] Bonjer HJ, Deijen CL, Haglind E; COLOR II Study Group. A Randomized Trial of Laparoscopic versus Open Surgery for Rectal Cancer. N Engl J Med. 2015 Jul 9;373(2):194. doi: 10.1056/NEJMc1505367. No abstract available. PMID 26154803
- [Background] Farges O, Goutte N, Bendersky N, Falissard B; ACHBT-French Hepatectomy Study Group. Incidence and risks of liver resection: an all-inclusive French nationwide study. Ann Surg. 2012 Nov;256(5):697-704; discussion 704-5. doi: 10.1097/SLA.0b013e31827241d5. PMID 23095612
- [Background] Tranchart H, Dagher I. Laparoscopic liver resection: a review. J Visc Surg. 2014 Apr;151(2):107-15. doi: 10.1016/j.jviscsurg.2013.10.003. Epub 2013 Dec 22. PMID 24365035
- [Background] Vigano L, Laurent A, Tayar C, Tomatis M, Ponti A, Cherqui D. The learning curve in laparoscopic liver resection: improved feasibility and reproducibility. Ann Surg. 2009 Nov;250(5):772-82. doi: 10.1097/SLA.0b013e3181bd93b2. PMID 19801926
- [Background] Castaing D, Vibert E, Ricca L, Azoulay D, Adam R, Gayet B. Oncologic results of laparoscopic versus open hepatectomy for colorectal liver metastases in two specialized centers. Ann Surg. 2009 Nov;250(5):849-55. doi: 10.1097/SLA.0b013e3181bcaf63. PMID 19801934
- [Background] Hasegawa Y, Nitta H, Sasaki A, Takahara T, Itabashi H, Katagiri H, Otsuka K, Nishizuka S, Wakabayashi G. Long-term outcomes of laparoscopic versus open liver resection for liver metastases from colorectal cancer: A comparative analysis of 168 consecutive cases at a single center. Surgery. 2015 Jun;157(6):1065-72. doi: 10.1016/j.surg.2015.01.017. Epub 2015 Mar 16. PMID 25791030
- [Background] Karagkounis G, Akyuz M, Guerron AD, Yazici P, Aucejo FN, Quintini C, Miller CM, Vogt DP, Fung JJ, Berber E. Perioperative and oncologic outcomes of minimally invasive liver resection for colorectal metastases: A case-control study of 130 patients. Surgery. 2016 Oct;160(4):1097-1103. doi: 10.1016/j.surg.2016.04.043. Epub 2016 Jul 30. PMID 27486002
- [Background] Schiffman SC, Kim KH, Tsung A, Marsh JW, Geller DA. Laparoscopic versus open liver resection for metastatic colorectal cancer: a metaanalysis of 610 patients. Surgery. 2015 Feb;157(2):211-22. doi: 10.1016/j.surg.2014.08.036. Epub 2014 Oct 1. PMID 25282529
- [Background] Tohme S, Goswami J, Han K, Chidi AP, Geller DA, Reddy S, Gleisner A, Tsung A. Minimally Invasive Resection of Colorectal Cancer Liver Metastases Leads to an Earlier Initiation of Chemotherapy Compared to Open Surgery. J Gastrointest Surg. 2015 Dec;19(12):2199-206. doi: 10.1007/s11605-015-2962-5. Epub 2015 Oct 5. PMID 26438480
- [Background] Topal H, Tiek J, Aerts R, Topal B. Outcome of laparoscopic major liver resection for colorectal metastases. Surg Endosc. 2012 Sep;26(9):2451-5. doi: 10.1007/s00464-012-2209-4. Epub 2012 Feb 23. PMID 22358126
- [Background] Polignano FM, Quyn AJ, Sanjay P, Henderson NA, Tait IS. Totally laparoscopic strategies for the management of colorectal cancer with synchronous liver metastasis. Surg Endosc. 2012 Sep;26(9):2571-8. doi: 10.1007/s00464-012-2235-2. Epub 2012 Mar 22. PMID 22437957
- [Background] Vanounou T, Steel JL, Nguyen KT, Tsung A, Marsh JW, Geller DA, Gamblin TC. Comparing the clinical and economic impact of laparoscopic versus open liver resection. Ann Surg Oncol. 2010 Apr;17(4):998-1009. doi: 10.1245/s10434-009-0839-0. Epub 2009 Dec 22. PMID 20033324
- [Background] Wakabayashi G, Cherqui D, Geller DA, Han HS, Kaneko H, Buell JF. Laparoscopic hepatectomy is theoretically better than open hepatectomy: preparing for the 2nd International Consensus Conference on Laparoscopic Liver Resection. J Hepatobiliary Pancreat Sci. 2014 Oct;21(10):723-31. doi: 10.1002/jhbp.139. Epub 2014 Aug 5. PMID 25130985
- [Background] Kazaryan AM, Marangos IP, Rosok BI, Rosseland AR, Villanger O, Fosse E, Mathisen O, Edwin B. Laparoscopic resection of colorectal liver metastases: surgical and long-term oncologic outcome. Ann Surg. 2010 Dec;252(6):1005-12. doi: 10.1097/SLA.0b013e3181f66954. PMID 21107111
- [Background] Makabe K, Nitta H, Takahara T, Hasegawa Y, Kanno S, Nishizuka S, Sasaki A, Wakabayashi G. Efficacy of occlusion of hepatic artery and risk of carbon dioxide gas embolism during laparoscopic hepatectomy in a pig model. J Hepatobiliary Pancreat Sci. 2014 Aug;21(8):592-8. doi: 10.1002/jhbp.103. Epub 2014 Apr 21. PMID 24753492
- [Background] Wu WC, Smith TS, Henderson WG, Eaton CB, Poses RM, Uttley G, Mor V, Sharma SC, Vezeridis M, Khuri SF, Friedmann PD. Operative blood loss, blood transfusion, and 30-day mortality in older patients after major noncardiac surgery. Ann Surg. 2010 Jul;252(1):11-7. doi: 10.1097/SLA.0b013e3181e3e43f. PMID 20505504
- [Background] Karakousis GC, Singer S, Zheng J, Gonen M, Coit D, DeMatteo RP, Strong VE. Laparoscopic versus open gastric resections for primary gastrointestinal stromal tumors (GISTs): a size-matched comparison. Ann Surg Oncol. 2011 Jun;18(6):1599-605. doi: 10.1245/s10434-010-1517-y. Epub 2011 Jan 5. PMID 21207158
- [Background] Pham TH, Perry KA, Dolan JP, Schipper P, Sukumar M, Sheppard BC, Hunter JG. Comparison of perioperative outcomes after combined thoracoscopic-laparoscopic esophagectomy and open Ivor-Lewis esophagectomy. Am J Surg. 2010 May;199(5):594-8. doi: 10.1016/j.amjsurg.2010.01.005. PMID 20466101
- [Background] Nobili C, Marzano E, Oussoultzoglou E, Rosso E, Addeo P, Bachellier P, Jaeck D, Pessaux P. Multivariate analysis of risk factors for pulmonary complications after hepatic resection. Ann Surg. 2012 Mar;255(3):540-50. doi: 10.1097/SLA.0b013e3182485857. PMID 22330041
- [Background] Lawrence VA, Cornell JE, Smetana GW; American College of Physicians. Strategies to reduce postoperative pulmonary complications after noncardiothoracic surgery: systematic review for the American College of Physicians. Ann Intern Med. 2006 Apr 18;144(8):596-608. doi: 10.7326/0003-4819-144-8-200604180-00011. PMID 16618957
- [Background] Soubrane O, Schwarz L, Cauchy F, Perotto LO, Brustia R, Bernard D, Scatton O. A Conceptual Technique for Laparoscopic Right Hepatectomy Based on Facts and Oncologic Principles: The Caudal Approach. Ann Surg. 2015 Jun;261(6):1226-31. doi: 10.1097/SLA.0000000000000737. PMID 24854453
- [Background] Fretland AA, Sokolov A, Postriganova N, Kazaryan AM, Pischke SE, Nilsson PH, Rognes IN, Bjornbeth BA, Fagerland MW, Mollnes TE, Edwin B. Inflammatory Response After Laparoscopic Versus Open Resection of Colorectal Liver Metastases: Data From the Oslo-CoMet Trial. Medicine (Baltimore). 2015 Oct;94(42):e1786. doi: 10.1097/MD.0000000000001786. PMID 26496309
- [Background] Veenhof AA, Vlug MS, van der Pas MH, Sietses C, van der Peet DL, de Lange-de Klerk ES, Bonjer HJ, Bemelman WA, Cuesta MA. Surgical stress response and postoperative immune function after laparoscopy or open surgery with fast track or standard perioperative care: a randomized trial. Ann Surg. 2012 Feb;255(2):216-21. doi: 10.1097/SLA.0b013e31824336e2. PMID 22241289
- [Background] Qiu J, Chen S, Pankaj P, Wu H. Laparoscopic hepatectomy is associated with considerably less morbidity and a long-term survival similar to that of the open procedure in patients with hepatic colorectal metastases. Surg Laparosc Endosc Percutan Tech. 2014 Dec;24(6):517-22. doi: 10.1097/SLE.0b013e31829cec2b. PMID 25187072
- [Background] Gigot JF, Glineur D, Santiago Azagra J, Goergen M, Ceuterick M, Morino M, Etienne J, Marescaux J, Mutter D, van Krunckelsven L, Descottes B, Valleix D, Lachachi F, Bertrand C, Mansvelt B, Hubens G, Saey JP, Schockmel R; Hepatobiliary and Pancreatic Section of the Royal Belgian Society of Surgery and the Belgian Group for Endoscopic Surgery. Laparoscopic liver resection for malignant liver tumors: preliminary results of a multicenter European study. Ann Surg. 2002 Jul;236(1):90-7. doi: 10.1097/00000658-200207000-00014. PMID 12131090
- [Background] Okunrintemi V, Gani F, Pawlik TM. National Trends in Postoperative Outcomes and Cost Comparing Minimally Invasive Versus Open Liver and Pancreatic Surgery. J Gastrointest Surg. 2016 Nov;20(11):1836-1843. doi: 10.1007/s11605-016-3267-z. Epub 2016 Sep 9. PMID 27613735
- [Background] Montalti R, Berardi G, Laurent S, Sebastiani S, Ferdinande L, Libbrecht LJ, Smeets P, Brescia A, Rogiers X, de Hemptinne B, Geboes K, Troisi RI. Laparoscopic liver resection compared to open approach in patients with colorectal liver metastases improves further resectability: Oncological outcomes of a case-control matched-pairs analysis. Eur J Surg Oncol. 2014 May;40(5):536-544. doi: 10.1016/j.ejso.2014.01.005. Epub 2014 Feb 2. PMID 24555996
- [Background] Nachmany I, Pencovich N, Zohar N, Ben-Yehuda A, Binyamin C, Goykhman Y, Lubezky N, Nakache R, Klausner JM. Laparoscopic versus open liver resection for metastatic colorectal cancer. Eur J Surg Oncol. 2015 Dec;41(12):1615-20. doi: 10.1016/j.ejso.2015.09.014. Epub 2015 Sep 30. PMID 26454765
- [Background] Ratti F, Catena M, Di Palo S, Staudacher C, Aldrighetti L. Impact of totally laparoscopic combined management of colorectal cancer with synchronous hepatic metastases on severity of complications: a propensity-score-based analysis. Surg Endosc. 2016 Nov;30(11):4934-4945. doi: 10.1007/s00464-016-4835-8. Epub 2016 Mar 4. PMID 26944725
- [Background] Allard MA, Cunha AS, Gayet B, Adam R, Goere D, Bachellier P, Azoulay D, Ayav A, Navarro F, Pessaux P; Colorectal Liver Metastases-French Study Group. Early and Long-term Oncological Outcomes After Laparoscopic Resection for Colorectal Liver Metastases: A Propensity Score-based Analysis. Ann Surg. 2015 Nov;262(5):794-802. doi: 10.1097/SLA.0000000000001475. PMID 26583668
- [Background] Cipriani F, Rawashdeh M, Stanton L, Armstrong T, Takhar A, Pearce NW, Primrose J, Abu Hilal M. Propensity score-based analysis of outcomes of laparoscopic versus open liver resection for colorectal metastases. Br J Surg. 2016 Oct;103(11):1504-12. doi: 10.1002/bjs.10211. Epub 2016 Aug 3. PMID 27484847
- [Background] Van Ness P. The concept of risk in biomedical research involving human subjects. Bioethics. 2001 Aug;15(4):364-70. doi: 10.1111/1467-8519.00244. PMID 11697390
- [Background] Tranchart H, Fuks D, Vigano L, Ferretti S, Paye F, Wakabayashi G, Ferrero A, Gayet B, Dagher I. Laparoscopic simultaneous resection of colorectal primary tumor and liver metastases: a propensity score matching analysis. Surg Endosc. 2016 May;30(5):1853-62. doi: 10.1007/s00464-015-4467-4. Epub 2015 Aug 15. PMID 26275554
- [Background] Untereiner X, Cagniet A, Memeo R, Tzedakis S, Piardi T, Severac F, Mutter D, Kianmanesh R, Marescaux J, Sommacale D, Pessaux P. Laparoscopic hepatectomy versus open hepatectomy for colorectal cancer liver metastases: comparative study with propensity score matching. Hepatobiliary Surg Nutr. 2016 Aug;5(4):290-9. doi: 10.21037/hbsn.2015.12.06. PMID 27500141
- [Background] Martinez-Cecilia D, Cipriani F, Shelat V, Ratti F, Tranchart H, Barkhatov L, Tomassini F, Montalti R, Halls M, Troisi RI, Dagher I, Aldrighetti L, Edwin B, Abu Hilal M. Laparoscopic Versus Open Liver Resection for Colorectal Metastases in Elderly and Octogenarian Patients: A Multicenter Propensity Score Based Analysis of Short- and Long-term Outcomes. Ann Surg. 2017 Jun;265(6):1192-1200. doi: 10.1097/SLA.0000000000002147. PMID 28151797
- [Background] Wong-Lun-Hing EM, van Dam RM, van Breukelen GJ, Tanis PJ, Ratti F, van Hillegersberg R, Slooter GD, de Wilt JH, Liem MS, de Boer MT, Klaase JM, Neumann UP, Aldrighetti LA, Dejong CH; ORANGE II Collaborative Group. Randomized clinical trial of open versus laparoscopic left lateral hepatic sectionectomy within an enhanced recovery after surgery programme (ORANGE II study). Br J Surg. 2017 Apr;104(5):525-535. doi: 10.1002/bjs.10438. Epub 2017 Jan 31. PMID 28138958
- [Background] Elshamy M, Takahashi H, Akyuz M, Yazici P, Yigitbas H, Hammad AY, Aucejo FN, Quintini C, Fung J, Berber E. Evolution of a laparoscopic liver resection program: an analysis of 203 cases. Surg Endosc. 2017 Oct;31(10):4150-4155. doi: 10.1007/s00464-017-5468-2. Epub 2017 Mar 31. PMID 28364151
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Nederlof N, Pessaux P, de Jonge J, Wijnhoven BP, Breitenstein S, Oberkofler CE, Graf R, Puhan MA, Clavien PA. The comprehensive complication index: a novel and more sensitive endpoint for assessing outcome and reducing sample size in randomized controlled trials. Ann Surg. 2014 Nov;260(5):757-62; discussion 762-3. doi: 10.1097/SLA.0000000000000948. PMID 25379846
- [Background] Balzan S, Belghiti J, Farges O, Ogata S, Sauvanet A, Delefosse D, Durand F. The "50-50 criteria" on postoperative day 5: an accurate predictor of liver failure and death after hepatectomy. Ann Surg. 2005 Dec;242(6):824-8, discussion 828-9. doi: 10.1097/01.sla.0000189131.90876.9e. PMID 16327492
- [Background] Ishizawa T, Hasegawa K, Kokudo N, Sano K, Imamura H, Beck Y, Sugawara Y, Makuuchi M. Risk factors and management of ascites after liver resection to treat hepatocellular carcinoma. Arch Surg. 2009 Jan;144(1):46-51. doi: 10.1001/archsurg.2008.511. PMID 19153324
- [Background] Koch M, Garden OJ, Padbury R, Rahbari NN, Adam R, Capussotti L, Fan ST, Yokoyama Y, Crawford M, Makuuchi M, Christophi C, Banting S, Brooke-Smith M, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Nimura Y, Figueras J, DeMatteo RP, Buchler MW, Weitz J. Bile leakage after hepatobiliary and pancreatic surgery: a definition and grading of severity by the International Study Group of Liver Surgery. Surgery. 2011 May;149(5):680-8. doi: 10.1016/j.surg.2010.12.002. Epub 2011 Feb 12. PMID 21316725
- [Background] Horan TC, Gaynes RP, Martone WJ, Jarvis WR, Emori TG. CDC definitions of nosocomial surgical site infections, 1992: a modification of CDC definitions of surgical wound infections. Am J Infect Control. 1992 Oct;20(5):271-4. doi: 10.1016/s0196-6553(05)80201-9. No abstract available. PMID 1332552
- [Background] Rahbari NN, Garden OJ, Padbury R, Maddern G, Koch M, Hugh TJ, Fan ST, Nimura Y, Figueras J, Vauthey JN, Rees M, Adam R, Dematteo RP, Greig P, Usatoff V, Banting S, Nagino M, Capussotti L, Yokoyama Y, Brooke-Smith M, Crawford M, Christophi C, Makuuchi M, Buchler MW, Weitz J. Post-hepatectomy haemorrhage: a definition and grading by the International Study Group of Liver Surgery (ISGLS). HPB (Oxford). 2011 Aug;13(8):528-35. doi: 10.1111/j.1477-2574.2011.00319.x. Epub 2011 Jun 7. PMID 21762295
- [Background] Cauchy F, Fuks D, Nomi T, Schwarz L, Barbier L, Dokmak S, Scatton O, Belghiti J, Soubrane O, Gayet B. Risk factors and consequences of conversion in laparoscopic major liver resection. Br J Surg. 2015 Jun;102(7):785-95. doi: 10.1002/bjs.9806. Epub 2015 Apr 2. PMID 25846843
- [Background] Blazeby JM, Fayers P, Conroy T, Sezer O, Ramage J, Rees M; European Organization for Research Treatment of Cancer (EORTC) Quality of Life Group. Validation of the European Organization for Research and Treatment of Cancer QLQ-LMC21 questionnaire for assessment of patient-reported outcomes during treatment of colorectal liver metastases. Br J Surg. 2009 Mar;96(3):291-8. doi: 10.1002/bjs.6471. PMID 19224519
- [Background] Graham JW, Olchowski AE, Gilreath TD. How many imputations are really needed? Some practical clarifications of multiple imputation theory. Prev Sci. 2007 Sep;8(3):206-13. doi: 10.1007/s11121-007-0070-9. Epub 2007 Jun 5. PMID 17549635